CLINICAL TRIAL: NCT02720237
Title: Reducing Hazardous Alcohol Use & Human Immunodeficiency Virus (HIV) Viral Load: A Randomized Controlled Trial (RCT) in Antiretroviral Therapy (ART) Clinics in Vietnam
Brief Title: Reducing Hazardous Alcohol Use & Human Immunodeficiency Virus (HIV) Viral Load
Acronym: REDART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Thai Nguyen Center for Preventive Medicine (Unknown); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0225b; 1R01DA037440-01 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-25 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Drinking; HIV
Keywords: Alcohol use; HIV; Viral Load; ART
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention; Motivational Interviewing; Methods; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief Intervention (Experimental): Brief Intervention (2 in-person sessions and 2 phone sessions), study assessment visits, and standard of care from providers at the ART clinic
  Interventions: Behavioral: Brief Intervention
- MET+CBT Intervention (Experimental): MET+CBT Intervention (6 in-person sessions and 3 optional group sessions), study assessment visits, and standard of care from providers at the ART clinic
  Interventions: Behavioral: Motivational Enhancement Therapy (MET) Intervention; Behavioral: Cognitive Behavioral Therapy (CBT) Intervention
- Assessment-Only Control (No Intervention): Study assessment visits and standard of care from providers at the ART clinic

INTERVENTIONS:
Behavioral: Brief Intervention — In-person individual sessions (occurring one month apart) and booster phone sessions (occurring 2-3 weeks after each in-person session), delivered by a trained counselor.
  Other Names: BI
  Arms: Brief Intervention
Behavioral: Motivational Enhancement Therapy (MET) Intervention — In-person individual sessions (one session per week) and optional group sessions, delivered by a trained counselor.
  Other Names: MET
  Arms: MET+CBT Intervention
Behavioral: Cognitive Behavioral Therapy (CBT) Intervention — In-person individual sessions (one session per week) and optional group sessions, delivered by a trained counselor.
  Other Names: CBT
  Arms: MET+CBT Intervention

SUMMARY:
The purpose of this study is to compare the effectiveness of two interventions [a Brief Intervention (BI) and a Motivational Enhancement Therapy+Cognitive Behavioral Therapy (MET+CBT) Intervention], against each other and with an assessment-only control, in improving both alcohol- and HIV-related outcomes, among hazardous and heavy drinking HIV-infected antiretroviral therapy (ART) clinic clients in Thai Nguyen, Vietnam.

DETAILED DESCRIPTION:
This study is a three-arm randomized controlled trial among hazardous and heavy drinking HIV-infected ART clinic clients in Thai Nguyen province, Vietnam. It compares the effects of two evidence-based, culturally adapted, behavioral interventions [a Brief Intervention (BI) and a Motivational Enhancement Therapy+Cognitive Behavioral Therapy (MET+CBT) Intervention] both against each other and compared with an assessment-only standard of care arm, in order to understand the relative effectiveness of each intervention in reducing alcohol use and suppressing HIV viral load.

The Brief Intervention (BI) consists of 2 individual sessions and 2 booster phone sessions delivered by a trained counselor and is based on Project Treat. Content of BI sessions includes review of drinking patterns, harmful effects of drinking, and alcohol use behavior change strategies. The MET+CBT Intervention consists of 6 sessions delivered by a trained counselor. The MET+CBT Intervention uses a client-centered, motivational interviewing approach and focuses on skills-building for alcohol use behavior change, including drinking refusal skills, skills to cope with and manage cravings and triggers, and developing positive thoughts and attitudes. It also includes review of drinking patterns and harmful effects of drinking.

This study will also measure the incremental cost-effectiveness of each intervention as compared to current counseling services offered in ART clinics in Vietnam.

Investigators hypothesize that: 1) Each intervention will be more effective than an assessment-only arm on percent days alcohol abstinent and percent virally suppressed at the 12-month assessment; 2) The BI will be equivalently effective to the MET+CBT Intervention on percent days alcohol abstinent; 3) The effect of each intervention on alcohol abstinence and viral suppression will be mediated by alcohol use readiness to change and/or coping skills acquisition; 4) The MET+CBT Intervention will be more effective than the BI on alcohol abstinence and viral suppression separately among participants with more severe alcohol use, people who inject drugs, and participants with depressive symptoms; 5) The alcohol reduction interventions (BI and MET+CBT Intervention) will be highly cost-effective compared to assessment-only standard of care; and 6) The BI will be highly cost-effective relative to the MET+CBT Intervention.

Understanding the relative effectiveness of each intervention in improving both alcohol- and HIV-related outcomes will provide insight into the optimal application of alcohol programs in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently a client on ART at the clinic
* Hazardous drinking, measured using the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) instrument: AUDIT-C score >= 4 for men, AUDIT-C score >=3 for women
* Plan on residing in Thai Nguyen province for the next 24 months

Exclusion Criteria:

* Unwilling to provide informed consent
* Unable to participate in study activities due to psychological disturbance, cognitive impairment or threatening behavior
* Unwilling to provide locator information
* Currently participating in other HIV, drug use or alcohol programs or interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Alcohol use | 12 months
  Percent days abstinent from alcohol
HIV viral load | 12 months
  Percent HIV viral suppression

SECONDARY OUTCOMES:
Number of participants who report a high level of readiness to change for alcohol use reduction | 12 months
  Readiness to change is assessed using a brief "Readiness to Change" questionnaire based on Rollnick et al. (1996), where response is captured using a 10-point Likert scale.
Number of participants who report a high level of coping skills for alcohol abstinence | 12 months
  Coping skills are assessed using the alcohol abstinence self-efficacy scale of DiClemente et al. (1994), where response is captured using a 10-point Likert scale.

OTHER OUTCOMES:
Cost-effectiveness of the alcohol reduction interventions | 3 months
  Assessed by the willingness-to-pay threshold of Vietnam's gross domestic product (GDP) per disability-adjusted life years (DALYs) averted
Health utility of the alcohol reduction interventions | 12 months
  Assessed using the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) instrument

CONTACTS AND LOCATIONS:
Overall Officials: Vivian F Go, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Thai Nguyen Center for Preventive Medicine, Thái Nguyên, Thai Nguyen, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JS, Hutton HE, Tran HV, Quang VN, Nguyen MX, Sripaipan T, Dowdy DW, Latkin CA, Chander G, Frangakis C, Go VF. Efficacy of Two Evidence-Based Alcohol Consumption Interventions on Positive, Negative, and Neutral Days Among Hazardous Alcohol Users Living with HIV in Vietnam. AIDS Behav. 2024 Feb;28(2):421-428. doi: 10.1007/s10461-023-04234-6. Epub 2023 Dec 12. PMID 38085428
- [Derived] Hershow RB, Reyes HLMN, Ha TV, Chander G, Mai NVT, Sripaipan T, Dowdy DW, Latkin C, Hutton HE, Pettifor A, Maman S, Frangakis C, Go VF. Evaluating the effects of two alcohol reduction counseling interventions on intimate partner violence perpetration: secondary analysis of a three-arm randomized controlled trial among Vietnamese men with HIV. Addiction. 2021 Oct;116(10):2712-2723. doi: 10.1111/add.15496. Epub 2021 Apr 27. PMID 33788329
- [Derived] Go VF, Hutton HE, Ha TV, Chander G, Latkin CA, Mai NVT, Quynh BX, Nguyen V, Sripaipan T, Lancaster KE, Blackburn N, Hershow RB, Dowdy DW, Frangakis C. Effect of 2 Integrated Interventions on Alcohol Abstinence and Viral Suppression Among Vietnamese Adults With Hazardous Alcohol Use and HIV: A Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2017115. doi: 10.1001/jamanetworkopen.2020.17115. PMID 32945875